CLINICAL TRIAL: NCT02463825
Title: A Registry-Based Randomized-Controlled, Double-Blinded Clinical Trial of Pimozide in Patients With Neuromuscular Junction Transmission Dysfunction Due to Amyotrophic Lateral Sclerosis
Brief Title: A Registry-Based Clinical Trial of Pimozide in Patients With Neuromuscular Junction Transmission Dysfunction Due to ALS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Collaborators: Hotchkiss Brain Institute, University of Calgary (Other)
Responsible Party: Principal Investigator, DR. LAWRENCE KORNGUT, Director, Calgary ALS and Motor Neuron Disease Clinic, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB14-0617
Record Dates: First submitted 2015-04-21; First posted 2015-06-04 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Pimozide; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 Pimozide (2mg per day) (Experimental): Pimozide will be initiated at 1 mg twice daily and maintained on 2mg/day for 50 days. End of study dose reduction will begin following the Final Outcome Measure Visit (Day 65). Pimozide will then be stopped.
  Interventions: Drug: Pimozide 2 mg per day
- Group 2 Pimozide (4mg per day) (Experimental): Pimozide will be initiated at 1 mg twice daily then increased by 1mg twice daily every five days to 4 mg/day) for 45 days. End of study dose reduction will begin following the Final Outcome Measure Visit (Day 65). Pimozide will be titrated by reducing the dose by 1 mg twice daily every day to full discontinuation (over 2 days).
  Interventions: Drug: Pimozide 4 mg per day
- Group 3 Placebo (Lactose tablet) (Placebo Comparator): Placebo tablets will be utilized and administered in an identical manner for subjects in Group 3
  Interventions: Drug: Placebo (Lactose tablet)

INTERVENTIONS:
Drug: Pimozide 2 mg per day
  Arms: Group 1 Pimozide (2mg per day)
Drug: Pimozide 4 mg per day
  Arms: Group 2 Pimozide (4mg per day)
Drug: Placebo (Lactose tablet)
  Arms: Group 3 Placebo (Lactose tablet)

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a neuromuscular disease that results in rapid decline in normal muscle function and tone leading to difficulties with mobility, eating, drinking, breathing, sleeping, and communicating. The disease is progressive and no cure currently exists. Most people diagnosed with ALS succumb within 3 to 5 years. The only approved treatment to slow the progression of ALS is called Rilutek® (riluzole) which has only a modest effect and has been shown to increase survival by a few months.

Muscular dysfunction present in people with ALS is caused by nerve breakdown and a dysfunction in the communication between the muscles and the nerves. The area where these communications occur is called the neuromuscular junction. Some recent studies have focused on using different medications to enhance communication at the neuromuscular junction with the goal of improving muscle function as a result. This approach is unproven but may help to slow the progression of the disease.

Pimozide is a medication that has been demonstrated to enhance communication at the neuromuscular junction in fish and mice. This study will look at whether Pimozide may help to slow the progression of ALS and how much medication needs to be taken to have an effect.

DETAILED DESCRIPTION:
This clinical trial has two components: an acute therapy component consisting of a Phase II placebo-controlled, double-blinded, randomized-controlled pilot study of pimozide for the treatment of ALS; and a second component featuring a longitudinal follow-up study on ALS progression and outcomes. This clinical trial is registry-based including subject recruitment facilitated by the Canadian Neuromuscular Disease Registry (CNDR; National Principal Investigator: L. Korngut), and longitudinal follow-up data collection will occur during the second component of this clinical trial through the CNDR.

The acute therapy study duration for each subject is around 11 weeks. The follow up study duration through the CNDR is up to 5 years.

Number of study participants:25

Randomization: Subjects will be block randomized with a block size of five subjects. Within each block one subject will be randomly assigned to placebo with the remaining four subjects randomized to the treatment groups. Study physicians will be blinded to patient randomization status. Randomization will occur with a 4:1 ratio of study drug (20 subjects) to placebo (5 subjects). After administration of maximum dose for 45-50 days, subjects will taper the allocated treatment or placebo. Randomization will occur via permuted block randomization and study personnel will be blinded to the randomization at all times allowing full concealment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients classified as having clinically definite, clinically probable, or clinically probable (laboratory-supported) ALS according to the El-Escorial diagnostic criteria for ALS
2. Evidence of decremental response greater or equal to 5.0% in at least one nerve-muscle pair at the initial screening visit
3. Age 18 years or greater
4. Consent to participate in the Canadian Neuromuscular Disease Registry (CNDR) (follow-up study component only).

Exclusion Criteria:

1. Diagnosis of clinically possible or clinically suspected ALS as defined by the El-Escorial diagnostic criteria for ALS
2. If the subject is taking riluzole the dose must be stable for 30 days prior to randomization visit. Riluzole cannot be initiated during the study.
3. History of Parkinson's disease
4. History of traumatic brain injury
5. History of neuroleptic malignant syndrome
6. History of hypersensitivity or serious adverse reaction(s) to a neuroleptic medication
7. History of prolonged QTc interval > 500 ms
8. History of hyponatremia < 130 mmol/L
9. History of current heparin or warfarin use
10. History of hepatic and/or renal impairment that may affect pimozide metabolism
11. History of current pregnancy or breastfeeding
12. Current antipsychotic use
13. Presence of central nervous system depression, comatose states, liver disorders, renal insufficiency, and blood dyscrasias
14. Presence of depressive disorders or Parkinson's syndrome
15. History of congenital long QT syndrome or with a family history of this syndrome and in patients with a history of cardiac arrhythmias or Torsade de Pointes
16. Presence of acquired long QT interval, such as associated with concomitant use of drugs known to prolong the QT interval
17. Presence of hypokalemia or hypomagnesemia
18. Presence of clinically significant bradycardia (heart rate < 50 beats per minute)
19. The concomitant use of CYP 3A4-inhibiting drugs such as azole antimycotics, antiviral protease inhibitors, macrolide antibiotics and nefazodone
20. The concomitant use of CYP 2D6-inhibiting drugs such as quinidine is also contraindicated
21. Concomitant use of serotonin reuptake inhibitors, such as, sertraline, paroxetine, citalopram and escitalopram
22. Severe dysphagia with risk of aspiration
23. Has taken any compound under current or known future study as a potential therapy for ALS less than 30 days prior to dosing OR history of exposure to stem cell therapy for treatment of ALS at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-08 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
ALS Functional Rating Scale-Revised (ALSFRS-R) | Change from randomization in ALSRSR-R at visit 5(day 51) and change from randomization in ALSFRS-R at visit 6 (day 65)
  A questionnaire based rating scale that assesses the functioning of ALS subjects across 4 domains: gross motor activity, fine motor activity, bulbar, and respiratory function
Slow Vital Capacity (SVC) | Change from screen (day -14) and randomization (day 1) in SVC at visit 5 (day 51), and Change from screen (day -14) and randomization (day 1) in SVC at visit 6 (day 65)
  SVC will be measured using a spirometer.
Decremental responses on repetitive nerve stimulation (DRRNS) | Change from screen (day -14) and randomization (day 1) in DRRNS at visit 5 (day 51), and Change from screen (day -14) and randomization (day 1) in DRRNS at visit 6 (day 65)
  Using Caldwell Electromyographic System, perform repetitive nerve stimulation studies and estimates of amplitude of decremental responses.

SECONDARY OUTCOMES:
Adverse Effects | Day 12, visit 3 (day 23), visit 4 (day 36), visit 5 (day 51), and visit 6 (day 65).
  Adverse event review will be conducted at study visits. Adverse events will be reported to the un-blinded study observer.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Korngut, MD, FRCPC, Principal Investigator — University of Calgary and Alberta Health Services
Locations (1):
- South Health Campus, Calgary, Alberta, Canada